CLINICAL TRIAL: NCT00143546
Title: Compassionate Use of Defibrotide for Patients With Veno-Occlusive Disease
Brief Title: Compassionate Use of Defibrotide for Patients With Veno-occlusive Disease of the Liver
Status: No longer available | Type: Expanded Access
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DETIDE
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Hepatic Veno-occlusive Disease
Keywords: Hepatic Veno-occlusive Disease
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — defibrotide

INTERVENTIONS:
Drug: Defibrotide — Defibrotide to be administered approximately every 6 hours at an initial dose of 6.25 mg/kg/dose. Subsequent doses will be escalated with a plateau of 15 mg/kg/dose (or 60 mg/kg/day total). For patients with persistent VOD, the dose may be escalated by 10 mg/kg/day as needed to a maximum of 110 mg/kg/day total.
  Other Names: Veno-occlusive disease; VOD; Hepatic veno-occlusive disease.

SUMMARY:
Veno-occlusive disease (VOD) of the liver is a significant complication for some patients undergoing hematopoietic stem cell transplantation. This disease is thought to be a toxicity secondary to chemotherapy or radiation-induced damage to the epithelial cells of the blood vessels in the liver. VOD is categorized as mild, moderate or severe. Historically, there has been no method to treat the disease. Recently, however, there have been investigations into the use of a new agent called defibrotide.

The primary purpose of this protocol is to provide defibrotide to patients with severe VOD. Because this drug has not been approved by the FDA, use of this medication under the auspices of this IND treatment plan is for compassionate use only.

DETAILED DESCRIPTION:
Secondary objectives of this protocol include the following:

* To describe the toxicities of defibrotide in patients with VOD.
* To describe the response rate of VOD in patients receiving defibrotide.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical or pathologic diagnosis of veno-occlusive disease. The following criteria will be used:

1. Hyperbilirubinemia (greater than or equal to 2mg/dl) and two of the following: (hepatomegaly, ascites, or weight gain [greater than or equal to 5% of baseline]); OR,
2. Patient who do not fulfill criteria in #1 but who have pathologic or radiographic evidence of VOD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-11

CONTACTS AND LOCATIONS:
Overall Officials: Wing Leung, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org